CLINICAL TRIAL: NCT05095233
Title: A Randomized Controlled Trial Targeting Intervention and Prevention of Suicide Risk (TIPS'r) Among University Students: CBT Vs Min Plan
Brief Title: MIN PLAN VS CBT for Suicide Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Syeda AYAT E ZAINAB Ali (Other)
Collaborators: Pakistan Institute of Living and Learning (Other); MinPlan Organization (Unknown)
Responsible Party: Sponsor-Investigator, Syeda AYAT E ZAINAB Ali, PhD Scholar, International Islamic University, Islamabad
Organization: International Islamic University, Islamabad (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LWL
Record Dates: First submitted 2021-09-11; First posted 2021-10-27 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Suicide Risk
Keywords: Suicidal ideation; Suicide Probability; Depression; CBT; Self Help Tool; MINPLAN
MeSH Terms: conditions — Suicidal Ideation; Depression | interventions — Psychosocial Intervention; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: The study is based on single blind randomized controlled trial with the randomization of study participants across two groups (1). Young Adults Culturally Adapted Manual Assisted Psychological Therapy (2). MINPLAN Tool
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Young Adults Culturally Adapted Therapy for Suicidal Prevention (Experimental): Young Adults Adapted Manual Assisted Psychological Therapy for Suicide Prevention
  Interventions: Behavioral: Young Adults Culturally Adapted Manual Assisted Psychological Therapy (YA-CMAP)
- MINPLAN TOOL (Active Comparator): Research has shown that user engagement, rather than the modality of therapy is the key to achieving successful outcomes and given that just 50% and 13% of patients currently have a choice of when and where they receive therapy, self-help tool apps Like MIN PLAN may not only be equally effective as some forms of traditional psychotherapy but also provide a flexible and pragmatic means of increasing patient access, through removing barriers to treatment that do not respond to financial impetus.
  Interventions: Device: Min Plan Tool

INTERVENTIONS:
Behavioral: Young Adults Culturally Adapted Manual Assisted Psychological Therapy (YA-CMAP) — YA-CMAP is a manual assisted brief psychological intervention based on the principles of Cognitive Behavior Therapy (CBT), including 8-10 sessions delivered over three months.
  This intervention includes evaluation of the suicide risk mainly suicidal ideation, psycho education, crisis skills, problem solving and simple cognitive techniques to manage emotions, negative thinking, relapse prevention strategies, training on interoceptive awareness, mood management and behavior.
  Other Names: Psychosocial Intervention; Cognitive Behavior Therapy
  Arms: Young Adults Culturally Adapted Therapy for Suicidal Prevention
Device: Min Plan Tool — Self-help Tool are common evidence-based methods to help deal with mental health problems.The 'MIN PLAN APP' aims to support people at risk of suicide by letting them create a safety plan based on cognitive therapeutic intervention and behavioral techniques.
  Arms: MINPLAN TOOL

SUMMARY:
1. To investigate the effectiveness of Young Adults Culturally Adapted Manual Assisted Psychological Therapy (YA-CMAP) in University students with Suicide Risk
2. To compare the effectiveness of Young Adults Culturally Adapted Manual Assisted Psychological Therapy (YA-CMAP) against MinPlan tool in University students with Suicide Risk

ELIGIBILITY:
Inclusion Criteria:

* Participants who are not taking any psychological help or psychotherapy in the past and present.
* Participants who are at risk of suicide without a history of suicidal attempts but with a history of suicidal ideation in the past two months will be included.

Exclusion Criteria:

* Participants with a history of substance misuse/drug dependence/alcohol dependence and psychosis.
* Participants diagnosed with dementia, schizophrenia, delirium, bipolar disorder, and learning disability.
* Participants with a diagnosis of DSM-V mental disorders due to general medical condition.
* Participants who are taking any psychiatric medication.
* Participants residing on a temporary basis in the study area.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Suicide Probability Scale | Assessments will be conducted at 3rd week after the baseline (1st follow up session), 6th week (2nd follow up session) and at 3rd month (3rd follow up session). Outcome assessment will be used to asses the change from baseline to follow-up.
  The Suicide Probability Scale (SPS) is a Likert-type scale which will be used to evaluate suicide probability in participants and consists of 36 items.
Suicidal Ideation | Assessments will be conducted at 3rd week after the baseline (1st follow up session), 6th week (2nd follow up session) and at 3rd month (3rd follow up session). Outcome assessment will be used to asses the change from baseline to follow-up.
  The Suicide Probability Scale (SPS) is a Likert-type scale with four subscales (hopelessness=12 items, suicide ideation=8 items, negative self evaluation=9 items and hostility=7 items), which has been developed by Cull and Wayne (1982). Suicidal Ideation will be measure through Suicide Probability Scale.

SECONDARY OUTCOMES:
Beck Depression Inventory-21 | Assessments will be conducted at 3rd week after the baseline (1st follow up session), 6th week (2nd follow up session) and at 3rd month (3rd follow up session). Outcome assessment will be used to asses the change from baseline to follow-up.
  Beck depression inventory-21 will be used to measure the symptoms of depression.
Psychache scale | Assessments will be conducted at 3rd week after the baseline (1st follow up session), 6th week (2nd follow up session) and at 3rd month (3rd follow up session).Outcome assessment will be used to asses the change from baseline to follow-up.
  Psychache scale is a 13-item scale that will be used to measures psychological/emotional or mental pain as conceptualized by Shneidman (1993).
Hopelessness | Assessments will be conducted at 3rd week after the baseline (1st follow up session), 6th week (2nd follow up session) and at 3rd month (3rd follow up session).Outcome assessment will be used to asses the change from baseline to follow-up.
  The Suicide Probability Scale (SPS) is a Likert-type scale with four subscales (hopelessness=12 items, suicide ideation=8 items, negative self evaluation=9 items and hostility=7 items), which has been developed by Cull and Wayne (1982). Hopelessness will be measure through Suicide Probability Scale.
Negative Self Evaluation | Assessments will be conducted at 3rd week after the baseline (1st follow up session), 6th week (2nd follow up session) and at 3rd month (3rd follow up session).Outcome assessment will be used to asses the change from baseline to follow-up.
  The Suicide Probability Scale (SPS) is a Likert-type scale with four subscales (hopelessness=12 items, suicide ideation=8 items, negative self evaluation=9 items and hostility=7 items), which has been developed by Cull and Wayne (1982). Negative Self Evaluation will be measure through SPS.
Hostility | Assessments will be conducted at 3rd week after the baseline (1st follow up session), 6th week (2nd follow up session) and at 3rd month (3rd follow up session).Outcome assessment will be used to asses the change from baseline to follow-up.
  The Suicide Probability Scale (SPS) is a Likert-type scale with four subscales (hopelessness=12 items, suicide ideation=8 items, negative self evaluation=9 items and hostility=7 items), which has been developed by Cull and Wayne (1982). Hostility will be measure through SPS.
Interpersonal Needs questionnaire | Assessments will be conducted at 3rd week after the baseline (1st follow up session), 6th week (2nd follow up session) and at 3rd month (3rd follow up session).Outcome assessment will be used to asses the change from baseline to follow-up.
  Interpersonal Needs questionnaire will be used to measure participants' beliefs about the extent to which they feel connected to others (i.e., belongingness) and the degree to which they feel they are a burden to others (i.e., burdensomeness).
Problem-Solving Inventory | Assessments will be conducted at 3rd week after the baseline (1st follow up session), 6th week (2nd follow up session) and at 3rd month (3rd follow up session).Outcome assessment will be used to asses the change from baseline to follow-up.
  The Problem-Solving Inventory is a 35-item instrument that measures perceptions of problem-solving behaviors and problem solving attitudes.
Multidimensional Assessment of Interoceptive Awareness (MAIA-2) | Assessments will be conducted at 3rd week after the baseline (1st follow up session), 6th week (2nd follow up session) and at 3rd month (3rd follow up session).Outcome assessment will be used to asses the change from baseline to follow-up.
  The Multidimensional Assessment of Interoceptive Awareness (MAIA-2) is an 8-scale state-trait questionnaire with 37 items to measure multiple dimensions of interoception by self-report.
Client Satisfaction Questionnaire (CSQ) | Assessments will be conducted at 3rd week after the baseline (1st follow up session), 6th week (2nd follow up session) and at 3rd month (3rd follow up session). This Questionnaire will be used to evaluate client satisfaction with mental health services.
  Client Satisfaction Questionnaire is a brief scale to measure the patient's satisfaction with mental health services.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Tamkeen Saleem, PhD, Study Chair — International Islamic University, Islamabad, Pakistan
Locations (1):
- International Islamic University, Islamabad, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Cognitive behavioral therapy approach for suicidal Thinking and behaviors in depression. — https://www.intechopen.com/chapters/41711